CLINICAL TRIAL: NCT03762577
Title: A Randomized Controlled Trial of Ground-based Walking Training for Adult Patients With Pulmonary Hypertension
Brief Title: Effects of Ground-based Walking Training in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozge Ertan, Physiotherapist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30146
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Walking Training; Exercise; Balance; Quality of Life
MeSH Terms: conditions — Hypertension, Pulmonary; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Training group will attend ground-based walking training under the supervision of a physiotherapist for 2 days and 30 minutes a week. Patients will walk for 1-2 days in a week without supervision.
  Interventions: Other: Ground-based walking training
- Control Group (No Intervention): Patient education will be given and no intervention will be made.

INTERVENTIONS:
Other: Ground-based walking training — Patients will attend a 2-day 30-minute ground-based walking training under the supervision of a physiotherapist. Patients will walk for 1-2 days in a week without supervision. According to the Modified Borg Scale, the dyspnea intensity will be 3-4 (medium to slightly difficult) and the heart rate will be completed to not exceed 120 min / pulse. Heart rate of patients will be followed by finger type pulse oximeter
  Arms: Training Group

SUMMARY:
Pulmonary Hypertension (PH) is a hemodynamic and physiopathological condition that is defined as an increase in pulmonary artery pressure ≥25 mmHg when measured at resting with symptoms such as dyspnea, fatigue, chest pain, and syncope. PH characterized by decreased exercise capacity, quality of life, peripheral muscle strength, balance, and physical inactivity. It is recommended that patients with PH should be included in cardiopulmonary rehabilitation programs in addition to medical treatment. Ground-based walking training is a safe and effective method for COPD patients. In the literature, there are no studies evaluating the effects of ground-based walking training in PH patients.

DETAILED DESCRIPTION:
The aim of this project is to determine the effect of ground-based walking training on physical activity, exercise capacity, balance, peripheral muscle strength and quality of life in patients with PH.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Diagnosed with PH
* Followed by the department of chest diseases at least six months
* Not participating in the rehabilitation program in last year

Exclusion Criteria:

* Functional group four due to WHO functional classification
* PH due to left heart diseases, PH due to lung diseases and/or hypoxia
* Treatment and medication change in the last three months
* Cooperation problems
* Patients with successful pulmonary endarterectomy operation
* Smoking
* Patients with uncontrolled cardiovascular diseases
* Patients with orthopeadic and/or neurologic disorders that could limit exercise tests
* Syncope history in recent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Endurance exercise capacity | 8 weeks
  endurance shuttle walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Ozge Ertan, Istanbul, Turkey (Türkiye)